CLINICAL TRIAL: NCT01141816
Title: Contrast-enhanced Ultrasound for Follow-up After Radiofrequency Ablation of Renal Lesions: a Prospective, Blinded Study
Brief Title: Contrast-enhanced Ultrasound for Follow-up After Radiofrequency Ablation of Kidney Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MIURCCCEUS
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cell carcinoma; radiofrequency ablation; contrast enhanced ultrasound; monitoring; follow up
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Masking Description: The radiologist is blinded to either CEUS or CT/MRI.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast-Enhanced Ultrasound (Experimental)
  Interventions: Other: Contrast-Enhanced Ultrasound

INTERVENTIONS:
Other: Contrast-Enhanced Ultrasound — Contrast-enhanced ultrasounds of the kidney will be performed within 7 days of routine CTs or MRIs at 3, 6, 12, 18, and 24 months post-radiofrequency ablation, with Perflutren Lipid Microsphere Injectible Suspension ('Definity') as the contrast agent.

SUMMARY:
Radiofrequency ablation (RFA) is an increasingly popular therapy option for treating small kidney cancer, especially for patients who are not ideal candidates for traditional surgery. Currently, follow-up after this procedure involves the patient having several CT scans (or MRI scans in some cases) over time to monitor for possible cancer recurrence. However, there are risks associated with the radiation exposure from CT scans and other risks, such as adverse events from the contrast media used in these scans. This study will therefore investigate whether a different technique, contrast-enhanced ultrasound (CEUS), can be an effective tool for follow-up monitoring of kidney cancer patients who have undergone RFA by comparing the results of their standard follow-up CT scans (or MRIs if applicable) with the results of CEUS. If CEUS is found to be just as effective as CT scans or MRIs in detecting kidney cancer recurrence, this technique could potentially become the new standard of care for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age and capable of giving informed consent
* patient undergoing CT of MRI for monitoring of renal lesions after radiofrequency ablation

Exclusion Criteria:

* pregnant patients
* patients with allergies to iodinated contrast agents
* patients with pulmonary hypertension, right-to-left cardiac shunts, or unstable cardiopulmonary disease (these are absolute or relative contraindications to the use of the ultrasound contrast agent, perflutren lipid microsphere)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity value of CEUS for tumour recurrence and by comparing to the standard CT/MRI. | 3 months post radiofrequency ablation procedure.
  The accuracy of contrast-enhanced ultrasound in monitoring renal lesions post-radiofrequency ablation will be assessed through sensitivity, specificity, and positive predictive value of CEUS for tumour recurrence and by comparing to the standard CT/ MRI.
Sensitivity value of CEUS for tumour recurrence and by comparing to the standard CT/MRI. | 6 months post radiofrequency ablation procedure.
  The accuracy of contrast-enhanced ultrasound in monitoring renal lesions post-radiofrequency ablation will be assessed through sensitivity, specificity, and positive predictive value of CEUS for tumour recurrence and by comparing to the standard CT/ MRI.
Sensitivity value of CEUS for tumour recurrence and by comparing to the standard CT/MRI. | 12 months post radiofrequency ablation procedure.
  The accuracy of contrast-enhanced ultrasound in monitoring renal lesions post-radiofrequency ablation will be assessed through sensitivity, specificity, and positive predictive value of CEUS for tumour recurrence and by comparing to the standard CT/ MRI.
Sensitivity value of CEUS for tumour recurrence and by comparing to the standard CT/MRI. | 18 months post radiofrequency ablation procedure.
  The accuracy of contrast-enhanced ultrasound in monitoring renal lesions post-radiofrequency ablation will be assessed through sensitivity, specificity, and positive predictive value of CEUS for tumour recurrence and by comparing to the standard CT/ MRI.
Sensitivity value of CEUS for tumour recurrence and by comparing to the standard CT/MRI. | 24 months post radiofrequency ablation procedure.
  The accuracy of contrast-enhanced ultrasound in monitoring renal lesions post-radiofrequency ablation will be assessed through sensitivity, specificity, and positive predictive value of CEUS for tumour recurrence and by comparing to the standard CT/ MRI.

SECONDARY OUTCOMES:
Quality of life data | 3 months post radiofrequency ablation
Quality of life data | 6 months post radiofrequency ablation
Quality of life data | 12 months post radiofrequency ablation
Quality of life data | 18 months post radiofrequency ablation
Quality of life data | 24 months post radiofrequency ablation

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada